CLINICAL TRIAL: NCT00950040
Title: Brief Alcohol Intervention to Reduce At-Risk Drinking Among Type 2 Diabetics
Acronym: SUGAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AA017418
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2016-04

CONDITIONS: At-risk Drinking; Type 2 Diabetes
Keywords: At-risk drinking; Type 2 diabetes; Treatment adherence; At-risk drinking among Type 2 diabetic patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Treatment Adherence and Compliance | interventions — Ethanol; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief alcohol intervention (Experimental): Brief alcohol intervention delivered in 2 15-minute in-person sessions and 2 5-minute telephone sessions.
  Interventions: Behavioral: Brief alcohol intervention
- General Health Education (Active Comparator): General health education intervention delivered in 2 15-minute in-person sessions and 2 5-minute telephone sessions.
  Interventions: Behavioral: General health education

INTERVENTIONS:
Behavioral: Brief alcohol intervention — The intervention consists of educational information, aspects of motivational interviewing, feedback concerning alcohol use and measures of glycemic control, alcohol use monitoring, and formulation of a change plan.
  Arms: Brief alcohol intervention
Behavioral: General health education — The intervention will consist of information about several general health behaviors.
  Arms: General Health Education

SUMMARY:
This study is designed to test an intervention to reduce at-risk drinking among Type 2 diabetic patients. At-risk drinking is associated with inferior diabetes treatment adherence and control. The investigators hypothesize that our brief alcohol intervention will result in a reduction in drinking and better diabetes treatment adherence and control. If successful, this intervention could help diabetics to gain better control of their diabetes and live healthier lives.

DETAILED DESCRIPTION:
At-risk drinking is common among diabetic patients and is associated with inferior diabetes treatment adherence and outcomes. While methods for reducing alcohol use in this population have been largely unexplored to date, brief interventions to reduce at-risk drinking have been well-validated in other patient populations and offer the promise to reduce at-risk drinking among diabetic patients, resulting in improved diabetes treatment adherence and outcomes.

We hypothesize that adding a brief alcohol intervention to standard diabetes treatment, relative to general health education, will reduce overall drinking volume and heavy drinking days among diabetic patients who are at-risk drinkers.

Furthermore, we expect participants who receive the brief alcohol intervention to have better diabetes treatment adherence and outcomes than the participants receiving general health education. We also expect that reduced alcohol consumption will mediate the effect of the brief alcohol intervention on diabetes treatment adherence and outcomes. In addition, we will explore potential treatment mechanisms.

The proposed study is a randomized, two-group design with repeated measures over time, comparing a brief alcohol intervention plus standard diabetes treatment to general health education. For this study, we will recruit a sample of 240 Type 2 diabetic patients from a large, urban primary care clinic. To be eligible for the study, patients must report at-risk drinking and poor diabetes treatment adherence.

This study holds the promise of establishing an efficacious intervention approach for Type 2 diabetic patients who are at-risk drinkers and are likely to maintain poor diabetes treatment adherence and outcomes in the absence of a change in their drinking behavior, resulting in increased diabetes-related morbidity and mortality. The intervention proposed in this study represents a novel approach to reducing at-risk drinking among diabetic patients that, if efficacious, can be readily integrated into the treatment of diabetes in a variety of treatment settings. In addition, this study will provide valuable information regarding the relationship between alcohol use and diabetes treatment adherence and outcomes and about the mechanisms of change in alcohol use among Type 2 diabetic patients who are at-risk drinkers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* have Type 2 diabetes,
* report at-risk drinking in past month,
* report poor diabetes treatment adherence.

Exclusion Criteria:

* current alcohol dependence or current psychoactive substance abuse or dependence (excluding nicotine),
* currently psychotic,
* unable to provide the name and contact information for a significant other to corroborate self-report,
* unable to provide the name and contact information for two people who could serve as locators, do not have access to a telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-07; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of drinks per day | 1, 3, 6, and 12 months
Percentage heavy drinking days | 1, 3, 6, and 12 months

SECONDARY OUTCOMES:
Summary of Diabetes Self-Care Activities subscale scores | 1, 3, 6, and 12 months
HbA1c levels | 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Ramsey, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States